CLINICAL TRIAL: NCT05194904
Title: Intrtavenous Ketorolac Versus Intravenous Dexmedetomidine for Postoperative Analgesia After Hypospadius Repair
Brief Title: Intravenous Dexmedetomidin on Postoperative Pain After Hypospadias Repair in Children
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Muhammed Samir Ghitany, resident, Assiut University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: intravenous dexmedetomidin
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Postoperative Pain
Keywords: dexmedetomidine; ketorolac
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; Ketorolac

STUDY DESIGN:
Intervention Model Description: This is a prospective randomised clinical study designed to assess the effect of intravenous ketorolac versus intravenous dexmedetomidin on postoperative pain after hypospadias repair in children
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 1 (Active Comparator): ketorolac group: number = 30 patients , time : after intubation, dose 0.9 mg/kg
  Interventions: Drug: Dexmedetomidine
- group 2 (Active Comparator): Dexmedetomidine group: number : 30 patients, time : after intubation, dose 1 μg/kg
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — This is a prospective randomised clinical study designed to assess the effect of intravenous ketorolac versus intravenous dexmedetomidin on postoperative pain after hypospadias repair in children
  Other Names: ketorolac

SUMMARY:
This study aimed to evaluate the efficacy of intravenous ketorolac versus dexmedetomidine as analgesia after Hypospadias repair surgery to determine the optimal procedure for pain control and postoperative reduction of analgesic use

DETAILED DESCRIPTION:
The guidelines of the American Society of Anesthesiologists (ASA) for the treatment of pain in the perioperative period define postoperative acute pain as pain present in surgical patients following the procedure.1 Almost 80% of patients undergoing surgery experience postoperative pain, and 80% of them reported moderate to severe pain intensity.2 Inadequate management of postoperative pain may lead to development of complications and prolonged recovery time with increased morbidity and mortality rates in adults.3,4 Although equivalent data for children are not available, this evidence warrants caution in pediatric population too. Appropriate treatment of postoperative pain contributes to shorter time of hospitalization, lower hospital costs, and increased level of patient satisfaction. There is enough evidence that an ineffective treatment of postoperative pain is in positive correlation with delayed wound healing, and the negative development of pain perception and chronic pain in the future.5,6 Hypospadias repair surgery is an invasive procedure whose postoperative phase is very painful.7 Pain management can be counted as an important step in all surgeries, especially in pediatric and neonatal surgical procedures. It has been reported that up to 40% of the children undergoing surgeries suffer from moderate to severe post-operative pain.8 In addition to the significance of post-operative pain management in the quality of life and satisfaction of the patients, it plays a great role in minimizing the complications and improving the surgery outcome in certain types of surgeries. In hypospadias surgery, post-operative pain results in manipulation of wounds and consequent infection, hemorrhage, and wound dehiscence.9 These complications cause significant preventable morbidities. Post-operative pain management also alleviates the local and systemic inflammation resulting in more favorable outcomes.10

Ketorolac is a non-steroidal anti-inflammatory drug (NSAID) that has an analgesic efficacy similar to commonly used opioids, and that recently has found wide acceptance in the treatment of postoperative pain in a variety of surgical procedures. Ketorolac is used for moderate pain relief; it may be used to treat severe pain when associated with opioids, reducing the opioid dose. The advantage of this association is the reduction of opioid side effects such as respiratory depression, pruritus, urinary retention, sedation and nausea . 11,12,13 Dexmedetomidine is a highly selective α2-adrenergic receptor agonist commonly used in neurosurgery . The advantages of dexmedetomidine include reducing perioperative catecholamine to maintain intraoperative hemodynamic stability and exerting the unique neuroprotective effects by inhibiting the release of glutamate, pro-apoptotic proteins, and pro-inflammatory cytokines. In addition, previous studies have shown that it can reduce sedative and opioid consumption and provide better analgesic effects with lesser concern for side effects than opioids

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I & II.
* Age between 2 years & 6 years old.
* Body weight below 30 Kg.

Exclusion Criteria:

* Any contraindications to any drug used
* patients refusal
* recurrent surgery

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Total analgesic consumption in the first 24 hours after surgery | first 24 hours
  Total analgesic consumption in the first 24 hours after surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gao J, Sun Z, Xiao Z, Du Q, Niu X, Wang G, Chang YW, Sun Y, Sun W, Lin A, Bresnahan JC, Maze M, Beattie MS, Pan JZ. Dexmedetomidine modulates neuroinflammation and improves outcome via alpha2-adrenergic receptor signaling after rat spinal cord injury. Br J Anaesth. 2019 Dec;123(6):827-838. doi: 10.1016/j.bja.2019.08.026. Epub 2019 Oct 14. PMID 31623841
- [Result] Blaise G, Roy WL. Postoperative pain relief after hypospadias repair in pediatric patients: regional analgesia versus systemic analgesics. Anesthesiology. 1986 Jul;65(1):84-6. doi: 10.1097/00000542-198607000-00016. No abstract available. PMID 3729064